CLINICAL TRIAL: NCT00572182
Title: A Phase I Study of MK-0752 in Pediatric Patients With Recurrent or Refractory CNS Malignancies
Brief Title: MK0752 in Treating Young Patients With Recurrent or Refractory CNS Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This Phase I study was permanently closed to patient accrual on February 23, 2011, due to the discontinuation of support from MERCK.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000578114; U01CA081457 (NIH); PBTC-024 (Other: Pediatric Brain Tumor Consortium); NCI-09-C-0112; NCT00923208 (obsolete NCT alias)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood brain stem glioma; childhood central nervous system germ cell tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; childhood high-grade cerebral astrocytoma; childhood choroid plexus tumor; childhood craniopharyngioma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; childhood oligodendroglioma; recurrent childhood pineoblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; childhood atypical teratoid/rhabdoid tumor; childhood spinal cord neoplasm; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood visual pathway and hypothalamic glioma; childhood grade III meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Choroid Plexus Neoplasms; Familial ependymoma; Medulloblastoma; Oligodendroglioma; Rhabdoid Tumor; Spinal Cord Neoplasms; Optic Nerve Glioma | interventions — 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MK-0752 — This is a dose escalation study. Patients may receive 150, 200, 260 or 325 mg/m2 orally for 3 consecutive days of every 7 days for 28 days (dosing regimen 1 - closed to accrual 2/23/2010) or 800, 1000, 1400, or 1800 mg/m2 orally once weekly for 28 days (1 course). In the absence of unacceptable toxicity or disease progression, treatment may continue for 6 courses.

SUMMARY:
RATIONALE: MK0752 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of MK0752 in treating young patients with recurrent or refractory CNS cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the maximum tolerated dose (MTD) and recommended phase II dose of MK0752 administered for 3 consecutive days of every 7 days in 28 day courses to young patients with recurrent or refractory CNS malignancies (Dosing regimen 1 - closed to accrual 2/23/2010).
* To estimate the MTD and recommend a phase II dose of MK0752 administered once weekly in 28 day courses to young patients with recurrent or refractory CNS malignancies (Dosing regimen 2).
* To compared the MK0752 systemic exposure attained with each dosage level on the different dosing regimens.

Secondary

* To characterize the pharmacokinetics of MK0752.
* To document and describe toxicities associated with MK0752.
* To preliminarily define the antitumor activity of MK0752 within the confines of a phase I setting.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral MK0752 once daily on days 1-3, 8-10, 15-17, and 22-24 (dosing regimen 1 - closed to accrual 2/23/2010) or days 1, 8, 15, and 22 (dosing regimen 2). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Treatment may be extended up to 19 courses if the patient is benefitting from the treatment.

Patients undergo blood sample collection periodically for pharmacokinetic studies.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary CNS tumor

  * Patients with intrinsic brain stem tumors do not require histologic verification, but must have radiographic evidence of progression
* Recurrent disease or refractory to standard therapy
* No histologically benign brain tumors (e.g., low-grade glioma)

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) or Lansky PS 60-100%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count ≥ 1,000/μL
* Platelet count ≥ 100,000/μL (unsupported)
* Hemoglobin ≥ 8 g/dL (RBC transfusions allowed)
* Creatinine clearance OR glomerular filtration rate ≥ 70 mL/min OR serum creatinine based on age as follows:

  * 0.8 mg/dL (≤ 5 years of age)
  * 1.0 mg/dL (> 5 to ≤ 10 years of age)
  * 1.2 mg/dL (> 10 to ≤ 15 years of age)
  * 1.5 mg/dL (> 15 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* ALT ≤ 2.5 times ULN for age
* Albumin ≥ 2.5 g/dL
* Sodium, potassium, magnesium, and calcium normal
* Patients with neurological deficits are eligible provided these deficits are stable for ≥ 2 weeks prior to study registration
* No clinically significant systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study therapy or would likely interfere with the study procedures or results
* No known hypersensitivity to MK0752

PRIOR CONCURRENT THERAPY:

* Recovered from the acute toxic effects of all prior therapy
* At least 3 weeks since prior myelosuppressive anticancer chemotherapy (6 weeks for nitrosoureas)
* At least 7 days since prior investigational or biologic agents

  * At least 3 weeks since prior investigational or biologic agents that have a prolonged half-life or for which the patient has experienced ≥ grade 2 myelosuppression in the treatment course preceding discontinuation of therapy
* At least 3 half lives since prior monoclonal antibody therapy
* At least 6 months since prior total body irradiation or craniospinal radiotherapy
* At least 6 weeks since other prior substantial bone marrow irradiation
* At least 2 weeks since prior local palliative radiotherapy (small volume)
* At least 6 months since prior allogeneic bone marrow transplantation (BMT)

  * No evidence of active graft versus host disease
* At least 3 months since prior autologous BMT or stem cell transplantation
* At least 7 days since prior hematopoietic growth factors (filgrastim [G-CSF], sargramostim [GM-CSF], or erythropoietin) (14 days for long-acting formulations)
* No prior MK0752
* No concurrent enzyme-inducing anticonvulsant drugs (EIACDs)
* No other concurrent anticancer or investigational drug therapy
* Concurrent dexamethasone allowed provided patient is on a stable or decreasing dose for ≥ 2 weeks prior to study registration

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | First 28 days of treatment
MK0752 systemic exposure | Day 1 of course 1
  Serial blood samples for pharmacokinetic studies of MK-0752 will be collected with the first dose of course 1 at pre-specified times.

SECONDARY OUTCOMES:
Pharmacokinetics | Day 1 of course 1
  Serial blood samples for pharmacokinetic studies of MK-0752 will be collected with the first dose of course 1 at pre-specified times.
Toxicity | From day 1 of treatment until off study
Objective response rate | End of courses 2, 4, 6 and at the end of treatment
  Brain imaging to assess tumor response to the treatment is performed at baseline, at the end of courses 2, 4, 6 and at the end of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (12):
- United States (12):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - NCI - Pediatric Oncology Branch, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington